CLINICAL TRIAL: NCT06233253
Title: A Brief Online Mindfulness-Based Intervention to Decrease Pre-Procedural Anxiety Before a First-Time Screening Colonoscopy: A Pilot Randomized Controlled Trial
Brief Title: Online Mindfulness-Based Intervention to Decrease Pre-Procedural Anxiety Before a First-Time Screening Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Mira Katz, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OSU-23136; NCI-2023-10496 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2024-01-08; First posted 2024-01-31 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Colorectal Carcinoma
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (usual care) (Active Comparator): Patients receive usual care prior to their scheduled screening colonoscopy.
  Interventions: Other: Best Practice; Other: Medical Chart Review; Other: Survey Administration
- Group II (online mindfulness intervention) (Experimental): Patients receive an online mindfulness intervention including infographics and 5-minute meditations QD for 5 days prior to their scheduled screening colonoscopy.
  Interventions: Other: Medical Chart Review; Behavioral: Online Mindfulness Meditation; Other: Survey Administration

INTERVENTIONS:
Other: Best Practice — Receive usual care
  Other Names: standard of care; standard therapy
  Arms: Group I (usual care)
Other: Medical Chart Review — Ancillary studies
  Other Names: Chart Review
Behavioral: Online Mindfulness Meditation — Receive an online mindfulness intervention
  Other Names: Online MBSR; Online Mindful Meditation; Online Mindfulness Relaxation; Online Mindfulness-Based Stress Reduction; Web-Based Mindfulness Meditation
  Arms: Group II (online mindfulness intervention)
Other: Survey Administration — Ancillary studies

SUMMARY:
This clinical trial tests how well an online mindfulness-based intervention (MBI) works to decrease anxiety in patients before a first-time screening colonoscopy. Elevated pre-procedural anxiety can affect patient outcomes including bowel preparation adherence and quality, the amount of sedation required, procedure time, patient satisfaction, cancellation or no-shows, and intention for future cancer screening. Mindfulness is a form of meditation that focuses on staying within the present moment to reduce anxiety. Previous research supports mindfulness practice among cancer survivors to decrease anxiety, fear of cancer re-occurrence, and to improve quality of life. Online MBIs have the potential to include targeted meditations and educational information designed to promote behavior change. This study may help researchers learn whether a mindfulness intervention works to decrease anxiety in patients before a first-time screening colonoscopy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To establish intervention feasibility and acceptability, and to collect preliminary efficacy data on a developed online mindfulness-based intervention (MBI) to reduce pre-procedural anxiety before a first-time screening colonoscopy compared to usual care.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: Patients receive usual care prior to their scheduled screening colonoscopy.

GROUP II: Patients receive an online mindfulness intervention including infographics and 5-minute meditations once daily (QD) for 5 days prior to their scheduled screening colonoscopy.

After completion of study intervention, patients are followed up 1-2 days post-colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be ages 45-75
* Patients must be at average risk for colorectal cancer (CRC)
* Patients must have scheduled their first-time screening colonoscopy as an outpatient at Ohio State University (OSU) at least 14 days in advance
* Patients must be able to speak and read English
* Patients must have daily access to a working telephone, email address, and internet connection
* Patients must provide consent

Exclusion Criteria:

* Previous colonoscopy
* Colonoscopy for diagnostic purposes
* Auditory or visual impairment that prevents internet use
* Previous cancer diagnosis (other than skin cancer)
* Previous diagnosis of a mental health disorder
* Current mental health treatment
* Family history of CRC
* Personal history of inflammatory bowel disease (ulcerative colitis or Crohn's disease)
* Confirmed or suspected hereditary CRC syndrome, such as familial adenomatous polyposis or Lynch syndrome

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-09-29 (Actual); Primary Completion 2024-07-12 (Actual); Study Completion 2024-07-12 (Actual)

PRIMARY OUTCOMES:
Retention rate (Feasibility) | Up to 4 weeks
  Feasibility will be assessed by the number of patients referred, number of participants recruited, and missing data from surveys and medical records. Feasibility will be achieved with a retention rate of 90% throughout the intervention. An independent samples t-test will be conducted to compare State-Trait Anxiety Inventory: State-Subscale (STAI-S) scores. Linear regression will be conducted to assess the difference when controlling for potential confounding variables of interest.
Satisfaction with the intervention (Acceptability) | At follow-up (1-2 days after the colonoscopy)
  Acceptability will be assessed by the number of intervention materials accessed and time to complete study activities (infographics, meditations, and surveys) via embedded REDCap metrics. Participants within the MBI group will also report meditation satisfaction and state mindfulness immediately after each meditation in addition to intervention satisfaction during the follow-up survey. Will report an average satisfaction score with the intervention >= 6.0, measured using a 7-point Likert scale. An independent samples t-test will be conducted to compare STAI-S scores. Linear regression will be conducted to assess the difference when controlling for potential confounding variables of interest.

SECONDARY OUTCOMES:
Colonoscopy nervousness | At pre-colonoscopy assessment
  Anxiety specific to the bowel prep and colonoscopy will be assessed using a visual analogue scale. Will be analyzed using t-test.
Mindfulness | At follow-up (1-2 days after the colonoscopy)
  Will measure the trait mindfulness using The Philadelphia Mindfulness Scale, a 20-item self-report with subscales of awareness and acceptance. Will be analyzed using t-test.
Mindfulness knowledge | At follow up (1-2 days after the colonoscopy)
  Will be assessed using a 5-item score about mindfulness. An independent samples t-test will be conducted to compare STAI-S scores.
Colorectal screening knowledge | At follow up (1-2 days after the colonoscopy)
  Will be assessed using a 5-item score about colorectal (CRC) screening. Will be analyzed using t-test.
Attitudes about CRC and CRC screening | At follow up (1-2 days after the colonoscopy)
  Will be self-reported and measured on a 5-point Likert scale. Will be analyzed using t-test.
Bowel prep adherence | At pre-colonoscopy assessment
  Will be self-reported and measured on a 5-point Likert scale. Will be analyzed using chi-square test.
Bowel prep difficulty | At pre-colonoscopy assessment
  Will be self-reported and measured on a 5-point Likert scale. Will be analyzed using t-test.
Bowel prep quality | Up to 4 weeks
  Will be measured using the Boston Bowel Preparation Scale or 5-point Likert scale and medical chart review. Will be analyzed using t-test.
Cancellation/no-show | At pre-colonoscopy assessment
  Will be measured by attendance. Will be analyzed using chi-square test.
Heart rate | Up to 4 weeks
  Will be measured in beats per minute using medical chart review. Will be analyzed using t-test.
Blood pressure | Up to 4 weeks
  Will be measured in millimeter of mercury using chart review at time of check-in (the first recorded) to the endoscopy suite holding area. Will be analyzed using t-test.
Sedative dose | Up to 4 weeks
  Will be measured in milligrams using chart review. Will be analyzed using t-test.
Procedural time | Up to 4 weeks
  Will be measured in minutes using medical chart review. Will be analyzed using t-test.
Cecal intubation time | At post-colonoscopy
  Will be measured in minutes using medical chart review. Will be analyzed using t-test.
Endoscopy suite time | Up to 4 weeks
  Will be measured in minutes using medical chart review. Will be analyzed using t-test.
Procedure satisfaction | At follow up (1-2 days after the colonoscopy)
  Will be self-reported and measured on a 5-point Likert scale. Will be analyzed using t-test.
Intent for future CRC screening | At follow up (1-2 days after the colonoscopy)
  Will be self-reported and measured on a 5-point Likert scale. Will be analyzed using t-test.

CONTACTS AND LOCATIONS:
Overall Officials: Katz, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu